CLINICAL TRIAL: NCT05247086
Title: Usefulness of Negative Pressure Therapy After Mesh Removal Due to Chronic Infection: a Multicentric, Prospective, Randomized Study.
Brief Title: Negative Pressure Therapy After Infected Mesh Removal.
Acronym: ICROMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ICROMA PROJECT
Record Dates: First submitted 2022-02-09; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Infection, Surgical Site
MeSH Terms: conditions — Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Convention closure (No Intervention): Conventional closure of the surgical wound after mesh removal surgery.
- Negative pressure therapy (Experimental): Negative pressure therapy of the surgical wound after mesh removal surgery.
  Interventions: Device: Negative pressure therapy

INTERVENTIONS:
Device: Negative pressure therapy — After surgical wound closure we will apply negative pressure therapy
  Arms: Negative pressure therapy

SUMMARY:
Chronic mesh infection mesh is a complication with leads to a long hospital stays, reoperation and admissions through emergency department. Surgical site infection (SSI) after removal are 58-72.7% depending on the published series. New therapeutic lines are needed in order to improve outcomes after surgery such as negative pressure therapy.

The main objective is to determine the SSI differences depending on the use of negative pressure therapy after infected mesh removal.

Material and methods: multicentric, prospective, randomized and an open comparative study. Patients will be selected sequentially n=94. Each selected patient will be randomized in two groups: conventional closure of the surgical wound vs. negative pressure therapy with a 30-day follow-up.

DETAILED DESCRIPTION:
The surgeon will not know the patient's arm of study before the operation. Once the wound will be closed, we will let know what kind of closure the patient will need. Negative pressure therapy will be the same in all patients, in order to mantain homogeneity.

We will set appointments each day while he is hospitalized, and after the discharge: at 7 (+/- 1) and 30 (+/- 5).

We will collect demographic data before and during surgery, as well as in the postoperative period, including appointments.

ELIGIBILITY:
Inclusion Criteria:

* Any gender, adult. Age minimum limits 18.
* Infected chronic mesh.
* Signing of informed consent.

Exclusion Criteria:

* Enterocutaneous fistula or enteroatmospheric fistula.
* Infected chronic mesh related to parastomal hernia.
* Patients who will no complete the follow-up period.
* Informed consent denial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  Differences between surgical site infection between conventional closure vs negative pressure therapy

IPD SHARING:
Plan to Share IPD: No
The protocol will be shared by internal email with other researchers, they should approve the protocol.